CLINICAL TRIAL: NCT05109975
Title: A Phase 1, Dose-finding Study of Debio 0123 as Monotherapy in Adult Patients With Advanced Solid Tumors, Followed by an Expansion Part to Assess Safety and Preliminary Anti-tumor Activity
Brief Title: A Study to Evaluate Safety and Preliminary Anti-tumor Activity of Debio 0123 as Monotherapy in Adult Participants With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Debio 0123-102; 2023-504824-24 (Other: EU CT number)
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Solid Tumors; WEE1-inhibitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Participants will receive Debio 0123 orally in escalating dose cohorts during each 21-day treatment cycle until progression of disease, unacceptable toxicity, participant's withdrawal, or Investigator's decision, whichever occurs first.
  Interventions: Drug: Debio 0123
- Part 2: Expansion (Experimental): Debio 0123 at the RP2D established in Part 1 participants with uterine serous carcinoma (USC) (arm A), recurrent or progressive, high-grade epithelial ovarian cancer (EOC) with cyclin E1 (arm B), and solid tumor with biomarker-driven selection (arm C).
  Interventions: Drug: Debio 0123

INTERVENTIONS:
Drug: Debio 0123 — Debio 0123 orally during 21-day treatment cycles.

SUMMARY:
This study has two parts: Part 1 and Part 2. The purpose of this study in Part 1, Dose Escalation Part is to determine the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of Debio 0123 as monotherapy with repeated dosing in adults with advanced solid tumors that recurred or progressed after prior therapy and/or for whom no standard therapy of proven benefit is available.

The purpose in Part 2, Expansion Part of this study, is to characterize the safety and tolerability of Debio 0123 in each study arm and overall when administered as monotherapy at the MTD/RP2D determined during the Dose Escalation Part 1 and to evaluate the preliminary anti-tumor activity of Debio 0123 when administered as monotherapy to participants in each study arm.

ELIGIBILITY:
Inclusion Criteria:

* Part 1 dose escalation only:

  * Histologically or cytologically confirmed locally advanced or metastatic solid tumors.
  * Measurable or non-measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria.
  * Disease progression under or following standard therapy and/or disease for which no available standard therapy of proven benefit.
* Part 2 expansion only:

  * Measurable disease per RECIST version 1.1 criteria for each arm.
  * Participants (≥18 years old) who progressed or have recurrence of one of the tumor types specified in the study arms following standard therapy according to RECIST version 1.1, or for whom, in the opinion of the Investigator, no effective standard therapy exists.
  * Arm A: Histologically or cytologically confirmed USC that recurred or progressed following at least 1 prior platinum-based line of therapy for management of advanced or metastatic disease.
  * Arm B: Histologically or cytologically confirmed, recurrent, high-grade EOC, primary peritoneal cancer, or fallopian tube cancer with cyclin E1 driven selection. Participants must have progressed after at least 1 prior platinum-based therapy for advanced/metastatic disease.
  * Arm C: Histologically or cytologically confirmed, locally advanced or metastatic solid tumor with biomarker-driven selection.
* Part 1 dose escalation and Part 2 expansion:

  * Accessible tumor for biopsy, and participant willing to undergo tumor biopsy unless archived tumor sample is available.
  * Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
  * Life expectancy of at least 3 months, in the best judgment of the Investigator.
  * Adequate bone marrow, liver biochemistry, renal function, and coagulation status.
  * Willing to practice highly effective methods of contraception.
  * Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Participants with active second malignancies requiring therapy in the last 6 months, with the exception of superficial bladder cancers, ductal carcinoma in situ or other carcinomas in situ, and non-melanoma non-melanoma skin cancers (basal cell/squamous cell skin cancer) that have been treated surgically.
* Current use of an investigational agent or a medical device.
* Major surgery ≤4 weeks prior to the first dose of study treatment or who have not recovered from the surgical procedure.
* Brain tumors and/or brain metastases unless they are asymptomatic, stable on recent imaging (not dated more than 28 days from the inclusion date), and have not required active treatment in the last month before study entry.
* History of myocardial infarction or stroke within 6 months, congestive heart failure greater than New York Heart Association (NYHA) class II, unstable angina pectoris, unexplained recurrent syncope, cardiac arrhythmia requiring treatment, family history of sudden death from cardiac-related causes before the age of 50, or any cardiotoxicity experienced after previous chemotherapy.
* Known infection requiring systemic use of an antibiotic or antiviral agent.
* Immunization with live or live-attenuated vaccine within 28 days prior to study inclusion or planned injection of live or live-attenuated vaccines.
* Pregnancy or breast-feeding.
* Inability or unwillingness to swallow oral medication.
* Clinically significant gastrointestinal abnormality that would affect the absorption of the drug.
* Any anti-cancer treatment, monoclonal antibodies/biologics, investigational treatment, or radiotherapy with curative intent within 28 days prior to starting study treatment. Palliative radiation for pain relief is allowed up to 1 week prior to starting study treatment.
* Unresolved AEs or toxicities due to previous treatments, i.e., >Grade 1. Exceptions will be made for Grade 2 anemia (if hemoglobin is not less than 9 g/dL or 5.6 mmol/L) and >Grade 2 alopecia and endocrinopathies controlled by replacement therapy (example, hypothyroidism due to immune checkpoint inhibitors).

[Note: Other inclusion/exclusion criteria mentioned in the protocol may apply.]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Part 1: Maximum Tolerated Dose (MTD) as Determined by Percentage of Participants with Dose Limiting Toxicities (DLTs) | Cycle 1 (each cycle is 21 days)
Part 1: Recommended Phase 2 Dose (RP2D) as Determined by Percentage of Participants with DLTs and Cumulative Safety Data | Cycle 1 (each cycle is 21 days)
Part 2: Percentage of Participants with Serious Adverse Events (SAEs) | Up to 30 days after the last dose of study treatment (up to 13 months)
Part 2: Percentage of Participants with Treatment-Emergent Adverse Events (TEAEs) and Laboratory Abnormalities | Up to 30 days after the last dose of study treatment (up to 13 months)
Part 2: Percentage of Participants with Treatment Discontinuations and Treatment Modifications due to Adverse Events (AEs) and Laboratory Abnormalities | Up to end of study treatment (up to 12 months)
Part 2: Overall Response Rate (ORR) | From the start of study treatment until disease progression (up to 12 months)

SECONDARY OUTCOMES:
Part 1: Percentage of Participants with SAEs | Up to 30 days after the last dose of study treatment (up to 13 months)
Part 1: Percentage of Participants with TEAEs and Laboratory Abnormalities | Up to 30 days after the last dose of study treatment (up to 13 months)
Part 1: Plasma Concentration of Debio 0123 | Pre-dose and at multiple time points up to 8 hours (h) on Day 1, Cycle 1 in Part 1 and 4 h on Day 1, Cycle 1 in Part 2 (each cycle is 21 days)
  The pharmacokinetics (PK) of Debio-0123 will be evaluated in plasma.
Parts 1 and 2: Anti-Tumor Activity as Assessed by Percentage of Participants with Tumor Response | Parts 1 and 2: Up to 12 months

CONTACTS AND LOCATIONS:
Locations (17):
- United States (4):
  - South Texas Accelerated Research Therapeutics (START) Midwest, Grand Rapids, Michigan
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Spain (9):
  - Hospital Universitario de A Coruna, A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Catala de Oncologia, Girona
  - Clinica Universidad de Navarra, Madrid
  - START Madrid. Hospital Fundación Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Clinico Universitario de Valencia, Valencia
- Switzerland (4):
  - Istituto Oncologico della Svizzera italiana - Ente Ospedaliero Cantonale, Bellinzona
  - Inselspital, Universitaetsspital Bern, Freiburgstrasse 4, Bern
  - Kantonsspital St. Gallen, Rorschacher Strasse 95, Sankt Gallen
  - Universitätsspital Zürich, Dermatologische Klinik, Zurich

IPD SHARING:
Plan to Share IPD: No